CLINICAL TRIAL: NCT06958003
Title: Neonatal Intensive Care Unit (NICU) Diaper Dermatitis: Prevention and Treatment With Airtime
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-091
Record Dates: First submitted 2025-04-21; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Diaper Dermatitis
MeSH Terms: conditions — Diaper Rash

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air Therapy (Experimental): Patients with receive 3-5 minutes of air therapy in addition to routine diaper care
  Interventions: Other: Air Therapy
- Routine Care (No Intervention): Patients will receive routine diaper care

INTERVENTIONS:
Other: Air Therapy — 3-5 minutes of air therapy in addition to routine diaper care
  Arms: Air Therapy

SUMMARY:
The purpose of this study is to investigate the use of 3-5 minutes air therapy for the prevention and treatment of diaper dermatitis in infants 30 weeks and older receiving care in the neonatal intensive care unit (NICU).

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at Good Samaritan Hospital NICU
* At least 30 weeks gestation at birth and corrected or older or corrected gestation
* Birth to 1 year old
* Stable vital signs (temperature, pulse, blood pressure, and oxygen saturation)

Exclusion Criteria:

* Parent/legal guardian unable or unavailable to consent to involvement in the study
* Congenital malformation impacting diaper area or spine

Ages: 30 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2025-01-21 (Actual); Primary Completion 2027-01-21 (Estimated); Study Completion 2027-04-21 (Estimated)

PRIMARY OUTCOMES:
Occurrence of diaper dermatitis | from admission to discharge from NICU, up to 6 months
  Whether infant is diagnosed with diaper dermatitis while in the NICU

CONTACTS AND LOCATIONS:
Overall Officials: Gina Marie Allaire, Principal Investigator — TriHealth Inc.
Locations (1):
- Good Samaritan Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No